CLINICAL TRIAL: NCT01733940
Title: Efficacy of Tegaderm-CHG® Dressing vs. Tegaderm-IV® Dressing in the Reduction of Central Catheter Colonization in Patients of the Intensive Care Unit of the University "Gómez Ulla" Hospital.
Brief Title: Efficacy of Tegaderm-CHG® Dressing vs. Tegaderm-IV® Dressing
Acronym: EAC-UCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Central de la Defensa Gómez Ulla (Other)
Responsible Party: Principal Investigator, ANA ISABEL LÓPEZ FIGUERAS, MD. Facultative of the Preventive Medicine Department, Hospital Central de la Defensa Gómez Ulla
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 10/12
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Intravascular Catheter Colonization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Tegaderm CHG" Dressing (Experimental): This arm is receiving a clorhexidine dressing for intravascular catheters.
  Interventions: Device: Application of a dressing with clorhexidine gluconate in intravascular catheters.
- "Tegaderm IV" dressing (Active Comparator): Use of tegaderm iv dressings for intravascular catheters. Change each 7 days.
  Interventions: Device: Application of a dressing without clorhexidine gluconate

INTERVENTIONS:
Device: Application of a dressing with clorhexidine gluconate in intravascular catheters.
  Arms: "Tegaderm CHG" Dressing
Device: Application of a dressing without clorhexidine gluconate
  Arms: "Tegaderm IV" dressing

SUMMARY:
Introduction: The vascular catheter-related bacteremia (BRC) is a major health problem in intensive care units. The use of dressings containing chlorhexidine gluconate (CHG) can decrease the catheters colonization, closely related to infection thereof.

Objective: To determine the efficacy of the dressing "Tegaderm CHG" dressings versus "Tegaderm IV" dressings in reducing the risk of colonization of central intravascular catheters in the intensive care unit (ICU).

Methods: Randomized controlled trial with blinding professional who reviews the main outcome. The study included patients over 18 years, indicating the central intravascular catheter implantation in the ICU or in the operating room, prior informed consent. Excluding subjects with positive blood culture at the time of catheter implantation.

The estimated sample size is 398 patients, with a confidence level of 95% and a statistical power of 80%. The study protocol was approved by the ethics committee of the hospital.

Be made prospectively followed subjects from study entry until catheter removal collecting information on age, sex, APACHEII, antibiotic therapy, duration of catheter insertion site and removal, reason for withdrawal and microbiological information.

For statistical analysis, a model is adjusted multivariate logistic regression, determining the interaction of variables with the likelihood ratio test and confusion by switching between the crude and adjusted effect greater than 10%.

Results and conclusions: The recruitment has started in November 2012 and is scheduled for completion in March 2013. This study will determine whether these new dressings are effective in our environment.

ELIGIBILITY:
Inclusion Criteria: over 18 years, indicating the central intravascular catheter implantation in the ICU or in the operating room, prior informed consent -

Exclusion Criteria:positive blood culture at the time of catheter implantation.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of intravascular central catheter colonization. | November 2012- March 2013

SECONDARY OUTCOMES:
Adverse effects of CHG Tegaderm ® dressings. | up to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital of the Defense, Madrid, Madrid, Spain